CLINICAL TRIAL: NCT00802815
Title: Double-blind, Randomized, Placebo-controlled Trial of Etanercept for 12 Months in Subjects With Inclusion Body Myositis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Glenn Lopate, Associate Professor of Neurology, Washington University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20031148
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Inclusion Body Myositis
MeSH Terms: conditions — Myositis, Inclusion Body | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept (Experimental)
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — 50 milligrams subcutaneously every week
  Other Names: Enbrel

SUMMARY:
Inclusion body myositis (IBM) is the most common late onset acquired muscle disease. Patients develop progressive weakness that may result in the need for assistive devices including a wheelchair. IBM may be due to abnormal immune activation, due in part to overproduction of tumor necrosis factor (TNF)-alpha. Etanercept blocks the activity of TNF-alpha, thereby blunting immune overactivation. Previous unblinded studies and case reports suggest that etanercept may improve strength or slow the progressive weakness in IBM. We are conducting a double-blind, randomized, placebo-controlled study to test if Etanercept is beneficial in slowing the progressive weakness in patients with IBM.

DETAILED DESCRIPTION:
Travel expenses not covered by the study.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of definite or probable IBM.
* Male or female aged 18-80.
* Subjects must be able to provide informed consent.
* Subjects must be on no immunosuppressive medication for 3 months and agree not to take immunosuppressive medication during the study.
* Subjects must not be on sulfasalazine
* Subjects or caregivers must be able to administer SQ medication.
* Women of childbearing potential (not postmenopausal or surgically sterile) must have a negative pregnancy test at screening and be using adequate birth control.
* Absence of exclusion criteria.

Exclusion Criteria:

* Exposure to etanercept within 3 months of study entry
* Exposure to other investigational drugs within 3 months of study entry.
* Subject with known hypersensitivity to etanercept.
* Subject with active medical or psychiatric condition that in the opinion of the principal investigator, may affect the interpretation of the safety and efficacy data or which otherwise contraindicates participation in the study.
* Signs, symptoms or laboratory evidence of severe renal, pulmonary, hepatic, neurologic, or cardiac (congestive heart failure, or coronary artery) disease, including creatinine > 2.0, LFT > 2x the upper limit of normal and hemoglobin < 12.5 (male) and < 11.0 (female).
* Subject with weakness from any other neurological or neuromuscular disease, including multiple sclerosis or other CNS demyelinating disease.
* Subject with sepsis or any active, chronic, or local infection or on antibiotic, antiviral or antifungal medication within 3 months prior to the first dose of Etanercept.
* A prior history of tuberculosis and/or a positive PPD skin test at screening (including reading of borderline, reactive but non-diagnostic) or prior inoculated subjects.
* Human immunodeficiency virus infection.
* Subject with history of opportunistic infection.
* Subject with a known history of anti-Jo-1, anti-SRP or anti-MI-2 antibodies.
* The presence of an associated connective tissue disease, including systemic lupus erythematous, Sjögren's syndrome, scleroderma or mixed connective tissue disease.
* History of a new diagnosis or treatment of invasive malignancy within 5 years of enrollment, including patients with a history of squamous cell carcinoma or basal cell carcinoma.
* History of drug or alcohol abuse within 1 year prior to study entry.
* Unwillingness to practice effective contraception, except for female patients who are post-menopausal or surgically sterile. The rhythm method is not to be used as the sloe method of contraception.
* Subjects are not to receive live vaccines while in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Quantitative Muscle Testing on 12 proximal and 12 distal muscles | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lopate, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Department of Neurology, St Louis, Missouri, United States